CLINICAL TRIAL: NCT06302842
Title: Pilot Open Label Study With Commercial Supplementation (Bioritmon Immuno Defend) in Healthy Subjects
Brief Title: Pilot Open Label Study With Commercial Supplementation in Healthy Subjects
Acronym: AUXNUTRIMMUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20J201
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Supportive Care
Keywords: Micronutrients; Innate immunity; Adaptive immunity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before and after treatment (Experimental): Nutraceutical (Bioritmon Immuno Defend), one oral preparation daily for 24 days.
  Immunological parameters are investigated before and after the treatment.
  Interventions: Dietary Supplement: Bioritmon Immuno Defend

INTERVENTIONS:
Dietary Supplement: Bioritmon Immuno Defend — Bioritmon Immuno Defend daily oral preparation for 24 days.

SUMMARY:
A bidirectional relationship among nutrition, infection and immunity exists: changes in one component affect the others. Various micronutrients are essential for immunocompetence, particularly vitamins A, C, D, E, B2, B6, and B12, folic acid, iron, selenium, and zinc. Micronutrient deficiencies are a recognized global public health issue, and poor nutritional status predisposes to certain infections. Immune function may be improved by restoring deficient micronutrients to recommended levels, thereby increasing resistance to infection and supporting faster recovery when infected. Diet alone may be insufficient and tailored micronutrient supplementation based on specific age-related needs is necessary.

Aim of the study is to investigate whether nutrient supplementation may affect different functional parameters of the innate and adaptive immunity.

DETAILED DESCRIPTION:
Study objective:

The study is designed to evaluate the effects of Bioritmon Immuno Defend on the immune response of healthy subjects.

The following parameters will be evaluated:

* PBMC proliferative response to polyclonal mitogens as described
* Expression of CD69 on mononuclear cells by flow cytometry before and after polyclonal stimulation as described
* Th1/Th2 cytokine cytoplasmic expression in PBMC before and after polyclonal stimulation
* Evaluation of NK cytotoxicity by NKTEST Tm BD Biosciences
* Evaluation of neutrophil phagocytic activity by PHAGOTESTTm BD Biosciences
* Evaluation of neutrophil oxidative burst by PHAGOBURST Tm BD Biosciences
* Evaluation of neutrophil chemotaxis by MIGRATEST Tm BD Biosciences
* Measurement of serum cytokines (IL2, IL4, IL6, IL10, IFNgamma, TNF) by solid phase assay as described

ELIGIBILITY:
Inclusion Criteria:

* Informed consent:
* Cooperative volunteers
* normal physical examination
* Female subjects: must not be pregnant, breastfeeding, or at risk to become pregnant during study participation. Female patients of childbearing potential, must test negative for pregnancy at the time of enrollment and agree to use a reliable method of birth control or remain abstinent during the study or for at least 30 days following the last dose of study drug, whichever is longer, or, must be a female of non-childbearing potential, defined as:
* women who have had surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation),
* women ≥60 years of age, or women ≥40 and <60 years of age who have had a cessation of menses for at least 12 months and a follicle-stimulating hormone (FSH) test confirming non-childbearing potential (FSH ≥40 mIU/mL).
* Have a negative COVID-19 antigen rapid test

Exclusion Criteria:

* Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study (i.e. Body Mass Index > 30, body temperature > 37,5°C)
* Diseases: Diabetes, cardiovascular, kidney, liver or lung diseases incompatible with exercise, active infections and cancer; angina pectoris or congestive heart failure in New York Heart Association class III-IV, severe chronic pulmonary disease, severe symptomatic obliterating arteriosclerosis, muscle- skeletal or cerebrovascular diseases incompatible with exercise training, drug or alcohol dependence and severe mental disease or any concurrent medical condition that, in the judgment of the PI, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being.
* Treatment with any investigational product (IP) during the study and within the 3 months (or at least 5 half-lives, whichever is longer) prior to Visit 1.
* Concomitant food supplements with Vitamins/lactoferrin or any other supplement, considered exclusionary by the PI and faculty physician, need to be avoided during the study.
* History of intolerance hypersensitivity or allergy to any of the component of the IP formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in neutrophil chemotaxis | Basal, after 12 and 24 days treatment
  Percentage increase of neutrophil chemotaxis
Change in neutrophil phagocytosis | Basal, after 12 and 24 days treatment
  Percentage increase of neutrophil phagocytosis
Change in neutrophil oxidative burst | Basal, after 12 and 24 days treatment
  Percentage increase of neutrophil oxidative burst
Change in mononuclear CD4pos69pos | Basal, after 12 and 24 days treatment
  Change in percentage of mononuclear CD4pos69pos
Change in mononuclear CD56pos69pos granzymepos | Basal, after 12 and 24 days treatment
  Change in percentage of mononuclear CD56pos69pos granzymepos
Change in plasma cytokine levels | Basal, after 12 and 24 days treatment
  Change in plasma cytokine levels (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Pier luigi Meroni, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No